CLINICAL TRIAL: NCT06009003
Title: Individual Patient Esmethadone (REL-1017) Expanded Access Program
Status: Temporarily not available | Type: Expanded Access
Sponsor: Relmada Therapeutics, Inc. (Industry)
Collaborators: Sponsor-Investigator (Unknown)
Responsible Party: Sponsor
Other Study IDs: REL-1017-EAP
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Depression
Keywords: REL-1017; esmethadone; Relmada; antidepressant; NMDA receptor antagonist; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: REL-1017 — REL-1017 tablet
  Other Names: esmethadone

SUMMARY:
To provide expanded access of esmethadone (REL-1017) to patients with a serious or immediately life-threatening disease or condition that may potentially benefit from esmethadone (REL-1017) who do not have access to other effective therapy and are not eligible for other clinical trials with esmethadone (REL-1017).

DETAILED DESCRIPTION:
The Expanded Access Program (EAP) is intended to provide pre-approval access to esmethadone (REL-1017) for eligible patients who suffer from a serious or immediately life-threatening disease or condition that may potentially benefit from esmethadone (REL-1017) as determined by the treating physician and have no satisfactory treatment options. This program is open in the United States and operates under the Individual Patient (also referred to as Single Patient) IND expanded access route in which the patient's treating physician serves as the sponsor. Expanded access requests must be from the patient's treating physicians and submitted according to the Relmada EAP policy at https://www.relmada.com/our-portfolio/eap.

ELIGIBILITY:
Inclusion Criteria:

* Patients who may potentially benefit from treatment with esmethadone (REL-1017) as determined by the treating physician.
* Have undergone appropriate standard treatments without success and in the opinion of the treating physician no comparable or satisfactory alternative treatment is available to treat the disease or condition.
* Are ineligible or unable to participate in any ongoing clinical study of the investigational product.
* Condition for which, in the opinion of the treating physician, there is sufficient evidence of a potential benefit from the use of the investigational product, and that potential benefit outweighs the known or anticipated risks.

Exclusion Criteria:

* History or presence of clinically significant health conditions which in the opinion of the Investigator would negatively impact the safety of the participant.
* History of QTc prolongation.
* History of allergy or hypersensitivity to methadone or related drugs.
* Pregnant or planning to become pregnant.
* Breast-feeding or planning to breast-feed.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Study Director — Relmada Therapeutics